CLINICAL TRIAL: NCT01973777
Title: A Pilot Study of Early Expulsion Rates of the IUB™ SCu380A Spherical Copper Intrauterine Contraceptive Device.
Brief Title: A Pilot Study of Early Expulsion Rates of the IUB™ SCu380A
Acronym: IUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wiebe, Ellen, M.D. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 130928 IUB
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Contraception
Keywords: intrauterine device, contraception

STUDY DESIGN:
Intervention Model Description: intrauterine contraceptive device IUB
Oversight: Data Monitoring Committee: No

ARMS (1):
- IUB (Experimental): There is one arm of women who will have IUBs inserted
  Interventions: Device: IUB

INTERVENTIONS:
Device: IUB — intrauterine contraceptive device
  Other Names: SCu380A IUB™

SUMMARY:
The IUB (Intrauterine ball) is a copper releasing intrauterine contraceptive device consisting of copper beads on a flexible NiTinol wire. It was designed to reduce the pain and bleeding caused by traditional T-shaped copper IUDs and to reduce expulsions. In an initial pilot of 15 women, there were no complications during the 12 months. This observational pilot study of 50 women will determine that the early expulsion rate is not greater than 10% and that there is patient and physician acceptance, so that we can plan a larger randomized controlled trial for efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* requesting non-hormonal intrauterine contraception
* able to return for ultrasound in 6-8 weeks

Exclusion Criteria:

* History of recent pelvic inflammatory disease
* Known anemia
* Dysfunctional uterine bleeding
* Malignancy or suspected malignant disease of female inner or outer genitalia
* Known intolerance or allergy to copper and/or copper IUDs
* Any other significant disease or condition that could interfere with the subject's ability to complete the protocol
* Pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Willow Women's Clinic, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- IUB Inserted: There is one arm of women who will have IUBs inserted
  IUB: intrauterine contraceptive device
Period: Overall Study
Arm/Group | IUB Inserted
Started | 51 (January 2014)
One Year Follow-up | 44
Completed | 44
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | IUB Inserted
Number analyzed (Participants) | 51
Age, Continuous [Mean (Full Range); unit: years] | 27 [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Expulsion Rate
Description: The device being expelled from the uterus as documented by ultrasound or by seeing the actual device outside the uterus
Time Frame: at 6-8 weeks
Measure: Number; unit: participants
Arm/Group | IUB Inserted
Number analyzed (Participants) | 49
participants | 9

2. Secondary Outcome: Complication
Description: infection, perforation, pregnancy
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | IUB Inserted
Number analyzed (Participants) | 44
participants | 1

3. Secondary Outcome: Acceptability
Description: patient-reported acceptability
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | IUB Inserted
Number analyzed (Participants) | 44
participants | 15

ADVERSE EVENTS:
Arm/Group | IUB Inserted
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 15/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IUB Inserted (N=51)
expulsions (Reproductive system and breast disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No